CLINICAL TRIAL: NCT01994226
Title: Multi-centre, Open-label, Active-comparator, Pragmatic Clinical Trial of Low-dose Colchicine Versus Naproxen in Patients With Acute Gout.
Brief Title: Colchicine Or Naproxen Treatment for ACute gouT
Acronym: CONTACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keele University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 149/11
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Colchicine; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose colchicine (Active Comparator): 500 mcg every eight hours for four days
  Interventions: Drug: Low-dose colchicine
- Naproxen (Active Comparator): Single initial dose of 750 mg followed by 250 mg every eight hours for up to seven days
  Interventions: Drug: Naproxen 750 mg/250 mg

INTERVENTIONS:
Drug: Low-dose colchicine — Route of Administration: Tablet - Oral Use
  Dose: 500 mcg (one tablet) every eight hours for four days
  Other Names: Colchicine 500 mcg
  Arms: Low-dose colchicine
Drug: Naproxen 750 mg/250 mg — Route of Administration: Tablet - Oral Use
  Dose: Single initial dose of 750 mg (three tablets) followed by 250 mg (one tablet) every eight hours for up to seven days
  Arms: Naproxen

SUMMARY:
Gout is the most common cause of inflamed joints affecting 1.4% of adults in the UK. Most patients are treated entirely in general practice yet primary care management is frequently suboptimal. Acute attacks of gout are excruciatingly painful and require urgent drug treatment to reduce inflammation, most commonly with antiinflammatory drugs(NSAIDs) or colchicine. In primary care, NSAIDs are most commonly used but can cause serious side effects such as stomach ulcers and heart disease, particularly in the elderly. Patients frequently require repeat prescriptions for recurrent attacks of acute gout increasing the risk of drug-related side-effects. Low-dose colchicine is popular amongst rheumatologists as it is effective and well tolerated. However, general practitioners (GPs) prescribe colchicine infrequently, probably because in the past the recommendation was for high doses to be prescribed which commonly caused severe diarrhoea. Recently, prescribing recommendations for colchicine have changed, advocating a lower dose regime.

Currently there is no evidence regarding whether NSAIDs or low-dose colchicine is the best treatment for acute gout. This trial will be the first direct comparison of the effectiveness and side effects of a NSAID (naproxen) and low-dose colchicine to treat acute gout in primary care. Naproxen will be used in this trial because it has been shown to be as effective as oral prednisolone for the treatment of acute gout, is safer than other commonly used NSAIDs such as diclofenac and indomethacin, and is inexpensive.

Patients consulting their GP with an acute attack of gout in up to 100 general practices will be invited to participate. Treatment success will be assessed by comparing pain reduction between the two drugs. The trial will also monitor side effects, quality of life, and cost effectiveness.

DETAILED DESCRIPTION:
Gout is the most prevalent inflammatory arthritis. It is largely managed in primary care but treatment is often suboptimal. Acute gout causes attacks of excruciating joint pain requiring rapid treatment. In primary care, treatment is most frequently with non-steroidal anti-inflammatory drugs (NSAIDs) which are effective but have frequent gastrointestinal, cardiovascular and renal side-effects, particularly in the elderly. Oral colchicine has been used to treat acute gout for many years although high-doses can cause intolerable gastrointestinal side-effects. Low-dose colchicine is thought to be as effective and better-tolerated and is now recommended by the British National Formulary. However, there has been no direct comparison of NSAID and low-dose colchicine for acute gout.

This pragmatic randomised trial will compare the effectiveness of low-dose colchicine (500 mcg three times every eight hours) and naproxen (750 mg immediately followed by 250 mg every eight hours) for reducing pain in adults aged 18 years and over consulting their GP with acute gout, recruited from up to 100 general practices. People experiencing their first attack of gout or a recurrent attack will be eligible to participate. However, all patients registered with each participating practice who have consulted with gout in the preceding two years will be mailed a letter of invitation and Participant Information Sheet informing them that the trial is taking place and encouraging them to consult their GP if they experience an attack of acute gout. Eligibility assessment, informed consent, randomisation, baseline data collection and prescription will be performed when the patient consults in primary care with acute gout. Outcome measures will be collected via self-complete questionnaires at days 1-7 (daily diary), and 4 weeks. The primary outcome measure will be change in worst pain intensity in the previous 24 hours measured daily over days 0-7. Secondary outcome measures include side-effects, time to treatment response, patient global assessment of response to treatment, adherence to treatment, use of other medications for pain relief, and cost. A sample size of 200 patients per treatment arm provides 90% power to detect a minimum clinically important treatment effect of a small standardised effect size of 0.3 between the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and over
* Consultation with GP, primary care out-of-hours service or walk-in-centre
* Current attack of acute gout (first attack or recurrent).
* Patient has capacity and willingness to give consent and complete the trial paperwork

Exclusion Criteria:

* Known unstable medical conditions (such as ischaemic heart disease, impaired liver function)
* Known stage 4/5 kidney disease (eGFR/creatinine clearance <30ml/min)
* Recent surgery or gastrointestinal bleed
* History of gastric ulcer
* Current anticoagulant use
* Allergy to aspirin/NSAID
* Previous inability to tolerate naproxen or low-dose colchicine
* Other contraindication to either study drug in accordance with the Summary of Product Characteristics (SPC)
* Prescription of naproxen or colchicine in the previous 24 hours
* Pregnant or lactating females
* Potentially vulnerable
* Previous participation in the CONTACT trial during a previous acute attack of gout.
* Involvement in another clinical trial of an investigational medicinal product in the last 90 days or any other research within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Roddy, Study Chair — Cheif Investigator
Locations (1):
- Keele University, Stoke-on-Trent, United Kingdom

REFERENCES:
- [Derived] McKenzie BJ, Wechalekar MD, Johnston RV, Schlesinger N, Buchbinder R. Colchicine for acute gout. Cochrane Database Syst Rev. 2021 Aug 26;8(8):CD006190. doi: 10.1002/14651858.CD006190.pub3. PMID 34438469
- [Derived] Roddy E, Clarkson K, Blagojevic-Bucknall M, Mehta R, Oppong R, Avery A, Hay EM, Heneghan C, Hartshorne L, Hooper J, Hughes G, Jowett S, Lewis M, Little P, McCartney K, Mahtani KR, Nunan D, Santer M, Williams S, Mallen CD. Open-label randomised pragmatic trial (CONTACT) comparing naproxen and low-dose colchicine for the treatment of gout flares in primary care. Ann Rheum Dis. 2020 Feb;79(2):276-284. doi: 10.1136/annrheumdis-2019-216154. Epub 2019 Oct 30. PMID 31666237

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-dose Colchicine: 500 mcg every eight hours for four days
  Low-dose colchicine: Route of Administration: Tablet - Oral Use
  Dose: 500 mcg (one tablet) every eight hours for four days
- Naproxen: Single initial dose of 750 mg followed by 250 mg every eight hours for up to seven days
  Naproxen 750 mg/250 mg: Route of Administration: Tablet - Oral Use
  Dose: Single initial dose of 750 mg (three tablets) followed by 250 mg (one tablet) every eight hours for up to seven days
Period: Overall Study
Arm/Group | Low-dose Colchicine | Naproxen
Started | 199 | 200
Completed | 180 | 179
Not Completed | 19 | 21
Not completed — Protocol Violation | 13 | 10
Not completed — Early Cessation of treatment | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Colchicine | Naproxen | Total
Number analyzed (Participants) | 199 | 200 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (13.4) | 58.7 (14.4) | 59.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 174 | 173 | 347
Region of Enrollment [Number; unit: participants]
  United Kingdom | 199 | 200 | 399

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: Worst pain intensity in last 24 hours using a 0 - 10 numeric rating scale, where high rates (10) indicate worst outcome
Time Frame: Days 0-7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low-dose Colchicine | Naproxen
Number analyzed (Participants) | 199 | 200
units on a scale | 3.5 (3.1) | 3.8 (3.2)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Low-dose Colchicine | Naproxen
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/200
Serious Adverse Events (participants affected / at risk) | 1/199 | 2/200
Other Adverse Events (participants affected / at risk) | 0/199 | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Colchicine (N=199) | Naproxen (N=200)
Non Cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Complication of TAVI procedure (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No